CLINICAL TRIAL: NCT01078844
Title: Memantine in Adult Autism Spectrum Disorder
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor withdrew funds
Sponsor: Johns Hopkins University (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NA_00015760
Record Dates: First submitted 2010-03-01; First posted 2010-03-02 (Estimated); Results first posted 2017-07-26 (Actual); Last update posted 2017-07-26 (Actual); Status verified 2017-06

CONDITIONS: Autism; Asperger's Disorder; Pervasive Developmental Disorder NOS
Keywords: Autism; Asperger's Disorder; Pervasive Developmental Disorder NOS; Adult; Memantine
MeSH Terms: conditions — Autistic Disorder; Asperger Syndrome; Child Development Disorders, Pervasive | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Treatment as usual plus placebo
  Interventions: Drug: Placebo
- memantine (Active Comparator): Treatment as usual plus memantine
  Interventions: Drug: memantine

INTERVENTIONS:
Drug: memantine — memantine 5-20 mg daily
  Arms: memantine
Drug: Placebo — Look-alike placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to see if memantine is helpful in managing problematic symptoms in adults with autism, Asperger's disorder, or Pervasive Developmental Disorder not otherwise specified (NOS).

ELIGIBILITY:
Inclusion criteria

* Participant is currently in treatment in the Johns Hopkins Bayview Medical Center (JHBMC)
* Participant has a diagnosis of:

  * Autistic Disorder
  * Asperger's Disorder
  * Pervasive Developmental Disorder (PDD) NOS
* Participant meets one of the following criteria:

  * CGI-S >= 4 (CGI-S: ________)
  * Participant has the following problematic behaviors (at least one) that might be expected to benefit from memantine:

    1. _____________________________________________
    2. _____________________________________________
    3. _____________________________________________

Exclusion criteria

The patient meets none of the following criteria (mark if absent):

* Active seizures (Patients with a history of seizures, who have been seizure-free on an antiepileptic regimen for six months or more would be eligible).
* Rett's Syndrome or Childhood Disintegrative Disorder
* Active treatment with an acetylcholinesterase inhibitor
* Prior or current treatment with memantine
* Current treatment with lamotrigine
* Genetic, metabolic or degenerative disorder (excepting Fragile X).
* Brain malformation or known severe brain trauma
* Pregnancy or breastfeeding
* Glomerular Filtration Rate (GFR) < 30 mL/min

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Samstad, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Brignell A, Marraffa C, Williams K, May T. Memantine for autism spectrum disorder. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013845. doi: 10.1002/14651858.CD013845.pub2. PMID 36006807

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 4 participants were enrolled in this study. It was terminated prematurely and the P.I. was never un-blinded. In an attempt to enter the information which was obtained within the confines of the system, all enrollment information and baseline characteristics have been entered into the experimental arm.
Groups:
- All Participants: Treatment as usual plus memantine
  memantine: memantine 5-20 mg daily
  OR
  Treatment as usual plus Placebo
Period: Overall Study
Arm/Group | All Participants
Started | 4
Completed | 0
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 4
Age, Customized [Count of Participants; unit: Participants]
  Age, years (18-85 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impression-Scale(CGI-S)
Time Frame: 12 weeks
Population: This study was terminated prematurely and data was not collected for this outcome measure.
Arm/Group | Placebo | Memantine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes